CLINICAL TRIAL: NCT07320911
Title: Patient-Specific Narrow-Slit Osteotomy Guides for Gap Arthroplasty in Pediatric TMJ Ankylosis
Brief Title: Patient-Specific Guides for Gap Pediatric Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-12-25/Artho-Tmj
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Ankylosis
Keywords: TMJ ankylosis; pediatrics; gap arthroplasty; CAD/CAM; surgical guide
MeSH Terms: conditions — Temporomandibular ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient-Specific Narrow-Slit Osteotomy Guides for Gap Arthroplasty (Experimental): Pediatric patient with TMJ Ankylosis managed with Patient-Specific Narrow-Slit Osteotomy Guides
  Interventions: Device: Patient-Specific Narrow-Slit Osteotomy Guides

INTERVENTIONS:
Device: Patient-Specific Narrow-Slit Osteotomy Guides — Patient-Specific Narrow-Slit Osteotomy Guides for gap arthroplasty

SUMMARY:
To date, few reports have combined patient-specific guides with piezoelectric devices for gap arthroplasty in children. This study evaluates the feasibility, accuracy, and early outcomes of this approach, hypothesizing that the combination of narrow-slit surgical guides and piezoelectric osteotomy provides safe and reproducible results in pediatric TMJ ankylosis.

DETAILED DESCRIPTION:
A prospective pilot study was conducted on [n] children (mean age [x] years) with TMJ ankylosis. Virtual surgical planning and CAD/CAM fabrication were used to design patient-specific guides with narrower osteotomy slits (width [x] mm) to allow precise bone removal and improved condylar fit. Preoperative and postoperative CT scans were superimposed to measure the accuracy of gap creation. Functional outcomes included maximal interincisal opening (MIO) at 1, 3, and 6 months, and complications.

ELIGIBILITY:
Inclusion Criteria:

1. patient with TMJ ankylosis.
2. less than 15 years old at the time of surgery

Exclusion Criteria:

1. Fibrous ankylosis without bony involvement
2. Associated craniofacial syndromes
3. Patients with systemic conditions contraindicating surgery

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
accuracy of the guide | 1 week
  Follow-up imaging was performed 1 week postoperatively using computed tomography (CT). Digital superimposition of the preoperative virtual plan and postoperative CT scans was carried out to assess the accuracy of osteotomy execution.

SECONDARY OUTCOMES:
mouth opening | 2 months
  inter-arch mouth opening assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study.